CLINICAL TRIAL: NCT00603174
Title: Use of Neurally Adjusted Ventilatory Assist in Infants With Acute Respiratory Failure: a Case Study on Servo I
Brief Title: Use of Neurally Adjusted Ventilatory Assist in Infants Respiratory Failure
Acronym: NAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Philippe Jouvet, Associate Professor, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJ 2537
Record Dates: First submitted 2007-11-21; First posted 2008-01-28 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Respiratory Failure
Keywords: NAVA; mechanical ventilation; infants; pediatric intensive care; infant
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Intubated and mechanically ventilated infants with respiratory failure (age < 1 year old). see inclusion-exclusion criteria.
  Interventions: Device: neurally adjusted ventilatory assist (NAVA)

INTERVENTIONS:
Device: neurally adjusted ventilatory assist (NAVA) — Following the titration of PEEP and the NAVA level, the infant will be ventilated on NAVA with the titrated levels. The following will be monitored and recorded for 20 min at 1 hour intervals: Phasic EAdi, tonic EAdi, tidal volume, ventilator-delivered pressure, respiratory rate, oxygen saturation, end tidal PCO2, and heart rate.

SUMMARY:
The present protocol will demonstrate the feasibility and efficacy of a newly developed mode of mechanical ventilation, Neurally Adjusted Ventilatory Assist, commonly known as NAVA. During NAVA, the timing and magnitude of pressure delivered are controlled by the infants' diaphragm electrical activity (EAdi), a validated measurement of neural respiratory drive. Recent clinical trials in adults and term infants have shown that NAVA is more synchronous than conventional pressure support ventilation, and that NAVA delivers lower mean airway pressures to achieve the same ventilation and respiratory muscle unloading. NAVA has recently been approved for use in infants by Health Canada and the FDA in the United States, and is commercially available on the Servoi ventilator (Maquet Critical Care, Solna, Sweden). The present protocol is designed as a "case study" where the researchers responsible would like to evaluate the feasibility and efficacy of ventilating an infant on NAVA with the Servoi for 12 hours, and to compare it to conventional ventilation.

DETAILED DESCRIPTION:
Research Design and Methods

Aim: To demonstrate the feasibility and efficacy of delivering NAVA in an intubated infant with the Servoi ventilator.

Measurements: All ventilatory and EAdi parameters will be stored in a laptop computer connected to the ventilator. SAO2 will be measured via pulse oximetry with a probe placed on one of the infant's extremities. End Tidal PCO2 measurements will also be made via probe placed on the Y piece of the respirator circuit.

General protocol sequence:

* All patients in the PICU at HSJ screened daily for eligibility
* Eligible cases reviewed with attending team and study team
* Informed consent obtained from parents or guardian
* Change to Servoi ventilator (conventional settings)
* Nasogastric tube replacement
* Monitor EAdi during conventional settings
* Adjust PEEP to minimize tonic activity
* NAVA level titration
* Application of NAVA for 12 hours with the titrated settings of PEEP and NAVA level.
* Return to conventional ventilator settings on servoi and monitor for 1 hour

NAVA for 12 hours Following the titration of PEEP and the NAVA level, the infant will be ventilated on NAVA with the titrated levels. The following will be monitored and recorded for 20 min at 1 hour intervals: Phasic EAdi, tonic EAdi, tidal volume, ventilator-delivered pressure, respiratory rate, oxygen saturation, end tidal PCO2, and heart rate.

The NAVA level and PEEP levels can be adjusted throughout the study period, and is based on clinical judgment (as they would routinely do for a conventional mode). Following any new setting, the 12 hour period will continue with those new settings. Following the end of this 12th hour of NAVA, the feeding tube with the sensors will remain in place for feeding the patient as per ICU protocol.

Protocol termination criteria: If the infant demonstrates a sustained change in any of the following, the protocol will be terminated:

* Sustained decrease in SaO2 < 92% requiring increase in FIO2 > 60%
* End tidal PCO2 > 60 mm Hg requiring progressive increases in the NAVA level,
* Sustained increase in heart rate>180 bpm during 15 min,
* Sustained increase in respiratory rate>60 bpm during 15 min,
* Uncontrolled agitation judged by the attending physician

Monitoring during conventional ventilation after discontinuation of NAVA (1 hour):

In order to compare NAVA to conventional ventilation, monitoring will be continued with conventional settings on the Servoi ventilator for 1 hour. The following will be monitored and recorded at 20 min intervals: Phasic EAdi, tonic EAdi, tidal volume, respiratory rate, saturation, CO2, HR. Following this, the baby will be returned to the ventilator and settings determined by the clinical team.

Primary outcomes:

* Patient-ventilator synchrony (trigger delays, cycling-off delays (Beck 2007))

Secondary outcomes:

* Phasic EAdi
* Tonic EAdi
* tidal volume, airway pressure, respiratory rate
* SAO2, End Tidal PCO2, FIO2 Number of times back-up rate started (per hour)
* Number of PEEP or NAVA level adjustments

Analysis and statistics

NAVA level titration: A continuous analysis will be performed breath-by-breath for phasic EAdi, ventilator-delivered pressure, respiratory rate and tidal volume. These values will be plotted versus the NAVA level. The NAVA level at the inflection point will be compared to the NAVA level initially used to match the conventional ventilation settings.

NAVA for 12 hours: EAdi signals will be processed automatically by the ventilator with standardized automated algorithms that have been implemented in to the Servoi. Phasic and tonic EAdi, as well as the ventilatory parameters (Vt, rr, SAO2, CO2) will be quantified breath-by breath and the last 20 min of each hour will be analyzed.

IN order to compare patient-ventilator synchrony between NAVA vs Conventional ventilation, trigger delays and cycling-off delays will be compared for each subject between the 2 modes. Paired t-tests will be used for this comparison.

Repeated measures ANOVA will be used to verify significant changes in variables over the twelve hour intervention period. The impact of PEEP on tonic diaphragm activity and the impact of NAVA level on tidal volume, pressures, and phasic diaphragm activity will also be compared by RM ANOVA.

Sample size determination: This is a case study and we will include 5 infants.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated infant with respiratory failure < 1 year old)
* Breathing spontaneously, as defined by the ability to trigger the ventilator
* The infant should be breathing on conventional ventilation (SIMV, assist control, or pressure support) with the following ventilator parameters: pressure plateau < 22 cm H2O (above PEEP) and PEEP ≤ 6 cm H2O.

Exclusion Criteria:

* Pneumothorax
* Degenerative neuromuscular disease
* Bleeding disorders
* Cardiovascular instability defined by vasopressors infusion (dopamine ≥ 5µg/kg/min, epinephrine, norepinephrine, dobutamine, vasopressin)
* Cyanotic congenital cardiovascular disease
* Phrenic nerve damage/diaphragm paralysis
* Esophageal perforation
* Use of high frequency oscillatory or jet ventilation
* Contraindication to changing naso gastric tube
* Infant is deemed "too unstable" by the attending physician

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
patient-ventilator synchrony | up to 28 days
  Patient-ventilator synchrony (trigger delays, cycling-off delays (Beck 2007))

SECONDARY OUTCOMES:
Tolerance | up to 28 days
  Evolution of tidal volume, airway pressure, respiratory rate, SAO2, End Tidal PCO2, FIO2
Number of times back-up rate started (per hour) in NAVA mode | up to 28 days
Number of PEEP or NAVA level adjustments in NAVA mode | up to 28 days
Phasic EAdi • Tonic EAdi Phasic EAdi and tonic EAdi | up to 28 days
  Phasic EAdi and tonic EAdi compared between pressure support, pressure control and NAVA modes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Jouvet, MD, Principal Investigator — Université de Montréal; Jennifer Beck, PhD, Principal Investigator — SunnyBrook Health Sciences Centre - Toronto
Locations (1):
- Research Center -CHU Sainte Justine - University of Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Sinderby C, Beck J, Spahija J, de Marchie M, Lacroix J, Navalesi P, Slutsky AS. Inspiratory muscle unloading by neurally adjusted ventilatory assist during maximal inspiratory efforts in healthy subjects. Chest. 2007 Mar;131(3):711-717. doi: 10.1378/chest.06-1909. PMID 17356084